CLINICAL TRIAL: NCT04980456
Title: Clinical Assessment of Two Daily Wear Monthly Replacement Soft Silicone Hydrogel Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLY935-C019
Record Dates: First submitted 2021-07-19; First posted 2021-07-28 (Actual); Results first posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-12

CONDITIONS: Myopia
Keywords: Contact lenses
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- TOTAL30, then Biofinity (Other): Lehfilcon A contact lenses worn first, followed by comfilcon A contact lenses as randomized. Each study product will be worn bilaterally (in both eyes) for approximately 30 days for at least 10 hours per day during waking hours only. CLEAR CARE will be used for daily cleaning and disinfection.
  Interventions: Device: Lehfilcon A contact lenses; Device: Comfilcon A contact lenses; Device: CLEAR CARE
- Biofinity, then TOTAL30 (Other): Comfilcon A contact lenses worn first, followed by lehfilcon A contact lenses, as randomized. Each study product will be worn bilaterally (in both eyes) for at least 10 hours per day during waking hours only. CLEAR CARE will be used for daily cleaning and disinfection.
  Interventions: Device: Lehfilcon A contact lenses; Device: Comfilcon A contact lenses; Device: CLEAR CARE

INTERVENTIONS:
Device: Lehfilcon A contact lenses — Investigational silicone hydrogel contact lenses
  Other Names: TOTAL30
Device: Comfilcon A contact lenses — Commercially available silicone hydrogel contact lenses
  Other Names: CooperVision® Biofinity®; Biofinity
Device: CLEAR CARE — Hydrogen peroxide-based cleaning and disinfecting solution

SUMMARY:
The purpose of this study is to compare the clinical performance of TOTAL30 contact lenses with Biofinity contact lenses over 30 days of daily wear.

DETAILED DESCRIPTION:
Subjects will wear two products and be expected to attend 4 office visits. The individual duration of participation will be approximately 65 days, which includes approximately 30 days of exposure to the test product and approximately 30 days of exposure to the comparator product.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign an approved Informed Consent form;
* Willing and able to attend all scheduled study visits as required by the protocol;
* Currently wearing any commercial spherical weekly/monthly soft contact lenses in both eyes for at least 3 months, minimum 5 days per week, 10 hours per day;
* Manifest cylinder less than or equal to 0.75 diopter (D) in each eye;
* Willing to stop wearing habitual contact lenses for the duration of study participation.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any eye condition that contraindicates contact lens wear, as determined by the Investigator;
* Any use of systemic or ocular medicine that contraindicates contact lens wear, as determined by the Investigator;
* Ocular or intraocular surgery (excluding placement of punctal plugs) within the previous 12 months or planned during the study;
* Any use of topical ocular medications and artificial tear or rewetting drops that would require instillation during contact lens wear;
* Current or prior Biofinity contact lens wear in the past 3 months prior to consent.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2021-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (14):
- United States (14):
  - Alcon Investigator 8135, Los Angeles, California
  - Alcon Investigator 8062, Oakland, California
  - Alcon Investigator 8106, San Francisco, California
  - Alcon Investigator 6356, Longwood, Florida
  - Alcon Investigator 6565, Maitland, Florida
  - Alcon Investigator 6654, West Palm Beach, Florida
  - Alcon Investigator 6567, Pittsburg, Kansas
  - Alcon Investigator 5582, Louisville, Kentucky
  - Alcon Investigator 8097, Sterling Heights, Michigan
  - Alcon Investigator 7980, Willmar, Minnesota
  - Alcon Investigator 8130, New York, New York
  - Alcon Investigator 6401, Warwick, Rhode Island
  - Alcon Investigator 6353, Memphis, Tennessee
  - Alcon Investigator 8175, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 14 investigative sites located in the United States.
Pre-assignment Details: Of the 257 enrolled, 8 subjects were exited prior to randomization as screen failures. This reporting group includes all subjects exposed to the study lenses, as treated (249). Note: One subject randomized to TOTAL30, then Biofinity was exposed to the incorrect study lenses in the sequence (Biofinity, then TOTAL30).
Units Other Than Participants: eyes
Groups:
- TOTAL30, Then Biofinity: Lehfilcon A contact lenses worn first, followed by comfilcon A contact lenses as randomized. Each study product was worn bilaterally (in both eyes) for approximately 30 days for at least 10 hours per day during waking hours only. CLEAR CARE was used for daily cleaning and disinfection.
- Biofinity, Then TOTAL30: Comfilcon A contact lenses worn first, followed by lehfilcon A contact lenses, as randomized. Each study product was worn bilaterally (in both eyes) for approximately 30 days for at least 10 hours per day during waking hours only. CLEAR CARE was used for daily cleaning and disinfection.
Period: Period 1 (Approximately 30 Days)
Arm/Group | TOTAL30, Then Biofinity | Biofinity, Then TOTAL30
Started | 122; 244 eyes | 127; 254 eyes
Completed | 119; 238 eyes | 124; 248 eyes
Not Completed | 3; 6 eyes | 3; 6 eyes
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2
Period: Period 2 (Approximately 30 Days)
Arm/Group | TOTAL30, Then Biofinity | Biofinity, Then TOTAL30
Started | 119; 238 eyes | 123; 246 eyes (One subject (2 eyes) discontinued after completing first period and prior to exposure to second period product due to an adverse event.)
Completed | 119; 238 eyes | 122; 244 eyes
Not Completed | 0; 0 eyes | 1; 2 eyes
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: All subjects exposed to any study lenses evaluated in this study, as randomized
Groups:
- TOTAL30, Then Biofinity: Lehfilcon A contact lenses worn first, followed by comfilcon A contact lenses, as randomized. Comfilcon A contact lenses worn first, followed by lehfilcon A contact lenses, as randomized. Each study product was worn bilaterally (in both eyes) for approximately 30 days for at least 10 hours per day during waking hours only. CLEAR CARE was used for daily cleaning and disinfection.
- Biofinity, Then TOTAL30: Comfilcon A contact lenses worn first, followed by lehfilcon A contact lenses, as randomized. Comfilcon A contact lenses worn first, followed by lehfilcon A contact lenses, as randomized. Each study product was worn bilaterally (in both eyes) for approximately 30 days for at least 10 hours per day during waking hours only. CLEAR CARE was used for daily cleaning and disinfection.
- Total: Total of all reporting groups
Arm/Group | TOTAL30, Then Biofinity | Biofinity, Then TOTAL30 | Total
Number analyzed (Participants) | 123 | 126 | 249
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.1 (7.7) | 33.1 (8.7) | 32.6 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 87 | 178
  Male | 32 | 39 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 8 | 17
  Not Hispanic or Latino | 114 | 118 | 232
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 80 | 79 | 159
  Black or African American | 4 | 5 | 9
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 37 | 41 | 78
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Other | 1 | 0 | 1
  Multi-racial | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 123 | 126 | 249

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean Distance VA (logMAR) With Study Lenses
Description: Distance visual acuity (VA) was assessed with study lenses in place. VA was collected for each eye separately using logarithmic of the Minimum Angle of Resolution (logMAR) charts. A logMAR acuity of 0.0 corresponds to 20/20 Snellen acuity (normal visual acuity), with a negative value denoting better than 20/20 visual acuity.
Time Frame: Day 30, each study product
Population: All subjects exposed to any study lenses evaluated in this study, as randomized, with non-missing response (eye)
Measure: Least Squares Mean (Standard Error); unit: logMAR
Units Other Than Participants: eyes
Groups:
- TOTAL30: Lehfilcon A contact lenses worn bilaterally (in both eyes) during Period 1 or Period 2, as randomized, for approximately 30 days at least 10 hours per day during waking hours only. CLEAR CARE was used for daily cleaning and disinfection.
- Biofinity: Comfilcon A contact lenses worn bilaterally (in both eyes) during Period 1 or Period 2, as randomized, for approximately 30 days at least 10 hours per day during waking hours only. CLEAR CARE was used for daily cleaning and disinfection.
Arm/Group | TOTAL30 | Biofinity
Number analyzed (Participants) | 240 | 243
Number analyzed (eyes) | 480 | 486
logMAR | -0.07 (0.005) | -0.08 (0.005)
Statistical Analysis 1: Comparison: TOTAL30 vs Biofinity; Test type: Non-Inferiority — Noninferiority in distance VA was declared if the least squares means difference upper confidence limit was less than 0.05; Since a noninferiority hypothesis is being tested, a p-value is not applicable. Confidence limit is being reported and compared to the noninferiority margin; Least Squares Mean Difference = 0.01, 95% CI 1-sided [upper limit 0.01], Standard Error of Mean 0.003 — LSM results based on mixed effects repeated measures model with both fixed (lens, visit, lens by visit interaction, period, and sequence) and random (subject) effects. Difference = TOTAL30 minus Biofinity

ADVERSE EVENTS:
Time Frame: Adverse events (AE's) were collected from time of consent to study exit, approximately 65 days.
Description: AE's were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of subjects. This analysis population includes all subjects/eyes exposed to any study lenses evaluated in this study
Groups:
- Pretreatment: Events reported in this group occurred prior to exposure to the study contact lenses
- TOTAL30 Ocular; TOTAL30 Nonocular: Events reported in this group occurred while exposed to the lehfilcon A contact lenses
- Biofinity Ocular; Biofinity Nonocular: Events reported in this group occurred while exposed to the comfilcon A contact lenses
Arm/Group | Pretreatment | TOTAL30 Ocular | TOTAL30 Nonocular | Biofinity Ocular | Biofinity Nonocular
All-Cause Mortality (participants affected / at risk) | 0/249 | 0/490 | 0/245 | 0/492 | 0/246
Serious Adverse Events (participants affected / at risk) | 0/249 | 0/490 | 2/245 | 0/492 | 0/246
Other Adverse Events (participants affected / at risk) | 0/249 | 0/490 | 0/245 | 0/492 | 0/246
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment (N=249) | TOTAL30 Ocular (N=490) | TOTAL30 Nonocular (N=245) | Biofinity Ocular (N=492) | Biofinity Nonocular (N=246)
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/56/NCT04980456/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/56/NCT04980456/SAP_001.pdf